CLINICAL TRIAL: NCT02217969
Title: Prospective, Randomized Trial of Alerting to Extended Hypotensive Exposures on Long-Term Outcome Following Adult Non-Cardiac Surgical Procedures: The SLUScore™ Trial
Brief Title: Prospective Trial of Alerting to Extended Hypotensive Exposures on Long-Term Outcome After Surgery
Acronym: SLUScore™
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB application withdrawn
Sponsor: St. Louis University (Other)
Responsible Party: Principal Investigator, Wolf H. Stapelfeldt, MD, Professor, St. Louis University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: IRB # 24886
Record Dates: First submitted 2014-08-13; First posted 2014-08-15 (Estimated); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia; Hypotension
Keywords: Anesthesia; Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electronic alert to SLUScore increase (Experimental): Patients whose anesthesia care team members are receiving alerts to increments in their SLUScore (progressive hypotensive exposures) are anticipated to be given interventions aimed at minimizing further hypotensive exposures. The decision of whether or not to intervene as well as the type(s) of interventions will be at the sole discretion of the patient's anesthesia care team
  Interventions: Behavioral: Electronic alert to SLUScore increase
- Control (no alert) (No Intervention): Routine anesthesia care at the discretion of the anesthesia care team

INTERVENTIONS:
Behavioral: Electronic alert to SLUScore increase — Treat hypotension to minimize further progression of the SLUScore
  Other Names: Treat hypotension
  Arms: Electronic alert to SLUScore increase

SUMMARY:
Patients undergoing anesthesia for non-cardiac surgery will be randomized to either having their anesthesia team alerted or kept blinded to extended periods of less than normal blood pressure with the goal of studying if providing these alerts leads to improved outcome after surgery (lower risk of death or complication in the days and weeks following surgery).

DETAILED DESCRIPTION:
Background:

We recently identified a significant association of postoperative morbidity and 30-day mortality with the concept of "hypotensive exposures" during anaesthesia. Specifically, we found in approximately 160,000 patients from 3 institutions (Cleveland Clinic, Vanderbilt University and Saint Louis University) that roughly every third adult patient undergoing a non-cardiac procedure under anaesthesia experienced twice the 30-day all-cause mortality portended by extended cumulative periods of less than normal intraoperative blood pressure. This association was independent of co-morbidity (Charlson Co-morbidity index), causing the same relative increase in mortality in "healthy" as in "sick" patients. A new method was introduced to quantify hypotensive exposures in form of a novel risk score called the SLUScore™, a score with values from ranging from 0 (no hypotensive exposure) to a maximum of 31 (the maximal number of exposures exceeded of a certain risk-based set of limits for time accumulated at a mean arterial blood pressure below thresholds between 75 and 45 mm Hg), with each increment of the SLUScore™ portending an equivalent 5% increase in 30-day postoperative mortality.

Hypothesis:

We test the hypothesis that alerting the anaesthesia care team to progressive hypotensive exposures (a progressive increase in their SLUScore™) improves 30-day survival. This will be tested in a prospective, randomised trial.

Methods and Design:

A novel Clinical Decision Support System (ACG-Anesthesia by Talis Clinical, LLC) will be used to alert anaesthesia care team members to patients' SLUScores™ in near real time (within 1 minute of documented exposures). At the time of transition from a SLUScore™ of 0 to 1 (occurring in approximately every third anaesthetic), patients will be automatically randomized by the ACG-Anesthesia system to either alert or no alert (blinded) status with the intent of raising awareness on the part of the anaesthesia care team in the alert group of the occurrence of extended hypotensive exposures and their associated risk, allowing the team to render its best clinical judgment to initiate interventions aimed at bringing patients out of progressive hypotensive states. With one interim analysis planned after two years, a total of 56,248 patients are projected to be enrolled over a 4-year period for this trial to be powered to detect a 0.3% absolute reduction in 30-day mortality, by saving at least 50 lives in the alert group after two years (two-sided p<0.016) or at least 70 lives (two-sided p<0.019) at the conclusion of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient presenting for any type of non-cardiac procedure performed under any type of anesthesia

Exclusion Criteria:

* Pediatric patients (< 18 yrs of age)
* Obstetric patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
30-day all-cause postoperative mortality | 30-days
  This addresses the known rather high rate of death within 30 days following non-cardiac surgical or interventional procedures

SECONDARY OUTCOMES:
Composite outcomes | one week
  Myocardial infarction; renal failure; septic shock

OTHER OUTCOMES:
Length of Hospital Stay | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Wolf H. Stapelfeldt, M.D., Principal Investigator — Saint Louis University School of Medicine
Locations (1):
- Saint Louis University Hospital, St Louis, Missouri, United States